CLINICAL TRIAL: NCT03775551
Title: Evaluation of the Effectiveness of an Improvement Collaborative Strategy to Improve the Counter-referral System of Patients With Cardiovascular Disease in the Public Healthcare Sector in Argentina
Brief Title: Counter-referral System Improvement Collaborative
Acronym: BIDCR-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Ministry of Public Health, Argentina (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C-RG-E1560-P002; 20180328 (Other: IECS)
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Quality Improvement
Keywords: quality improvement; collaborative; counter reference
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The participants belonging to the hospitals assigned to the control group the health providers will give feedback on their health condition and will advise on how to follow up their care after discharge or referral back to PHC following usual practice.
- Improvement cycle (Experimental): In participants belonging to the hospitals assigned to the intervention group,the health providers will give feedback on their health condition and will advise on how to follow up their care after discharge or referral back to PHC using innovative intervention to assure continuity of care and assistant level approach. This innovations will be crafted from the rapid improvement cycles considering the environment and key aspects of the every day care at the participating centers.
  Interventions: Behavioral: Improvement cycle

INTERVENTIONS:
Behavioral: Improvement cycle — at least 6 workshops (sessions) will be held with the members of the care system, in order to identify opportunities for improvement oriented to the design and application of an innovative intervention based on best practices.
  Other Names: quality improvement cycle
  Arms: Improvement cycle

SUMMARY:
Coordination between different levels of care has been identified as one of the main components of care among people with chronic diseases. In this sense, an adequate referral and counter-reference system facilitates the management of the care process with timely access to the required referral. The objective of this project is to evaluate the effectiveness of a multicomponent strategy that improves the counter- referral process in patients with cardiovascular diseases in the public health system.

Population: The study will be carried out in selected hospitals of the provinces of Mendoza, Tucumán and Salta in Argentina. Patients who have been hospitalized with a diagnosis of heart failure, hypertension (requires hospitalization) and / or coronary disease (unstable angina) will be included.

Design and methods: a Randomized clinical study by clusters. 10 hospital will be included: 5 will be randomly assigned to receive an intervention to increase the improve counter referral rates (improvement cycles) and 5 to the control branch (usual care). 51 participants will be included in each hospital, in total, 510 participants.

Intervention: An innovative vision is proposed, which combines a participatory and dynamic methodology based on improvement cycles. This approach includes the implementation of participatory learning sessions for health providers, involving the effectors of the design of the intervention. In the intervention branch at least 6 workshops (sessions) will be held with the members of the care system, in order to identify opportunities for improvement oriented to the design and application of an innovative intervention based on best practices. Each one of the sessions will constitute an analysis of the improvement cycle, following the following steps: 1) Selection of participants of the initial workshop; 2) Development of work model based on bibliographic review and initial qualitative phase; 3) Initial workshop with effectors for training in continuous improvement, objectives, interventions and data collection; 4) Learning workshops to discuss results, applicability of interventions and modifications to the work plan; 5) Closing session to evaluate preliminary results and discuss continuity of interventions beyond the project.

Outcomes: 1) consultation in the PHC after hospital discharge; 2) readmission's; 3) consultations in the hospital; 4) follow-up in the PHC; 5) patient perspective (satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Subjects that only have public health coverage or PAMI
* Adults over 18 year of age
* Patients admitted to the hospital with diagnosis of: non valvular heart failure and/or complicated hypertension ( that requires hospitalization) and/or coronary heart disease ( unstable angina)
* Residence in the area of influence of the hospitals

Exclusion Criteria:

* Pregnant women
* Anticoagulated patients
* People who are immobilized
* People who do not give their informed consent
* People who plan to move in the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Patients visits in a primary health center (PHC) after hospital discharge | 3 months after enrollment and/or end of study
  proportion of visits made in a primary care center (PHC) after hospital discharge

SECONDARY OUTCOMES:
Effective counter reference performed by physicians | 3 months after enrollment and/or end of study
  proportion of documented ( written) counter references by hospital physicians to a PHC
Time to the first consultation in a PHC after the hospital discharge | 3 months after enrollment and/or .end of study
  mean number of days upon patient hospital discharged to the first visit in a primary care center
Cardiovascular hospital readmission's | 3 months after enrollment and/or end of study
  proportion of re-admissions for the same primary admission condition for which the patient was discharged within the first 90 days
Cardiovascular re consultations at the second level of care | 3 months after enrollment and/or end of study
  proportions of cardiovascular consultations at the secondary level of care after hospital discharge that should have been performed at the first level of care related to the condition for which the patient was included and admitted to the hospital
Patients satisfaction with the primary health level measured by adapted PCAT questions | 4 months
  patients satisfaction with the health care provided at the PHC measured by adapted PTCA questions. The Primary Care Assessment Tool was design to evaluate attainment of features in primary care settings. Attributes identified by the tool are first contact accessibility and use, continuity, and coordination in the primary level. The tool has been adapted and validated in several countries and settings. The global index for evaluation will be composed as the sum of 10 items, ranging from 10 to 40. To facilitate interpretation the score will be transformed to a scale of 0 -100 points ( score =100 x (sum -10)/40-10), with higher score indicating more favorable satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Irazola, MD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy; Ezequiel García Elorrio, PhD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy
Locations (10):
- Argentina (10):
  - Hospital A Italo Perrupato, San Martín, Mendoza Province
  - Hospital Teodoro J. Schestakow, San Rafael, Mendoza Province
  - Hospital Antonio J. Scaravelli, Tunuyán, Mendoza Province
  - Hospital N. Joaquín Castellano, General Güemes, Salta Province
  - Hospital Centro de Salud Zenón J. Santillán, San Miguel de Tucumán, Tucumán Province
  - Hospital Ángel C. Padilla, San Miguel de Tucumán, Tucumán Province
  - Hospital Central, Mendoza
  - Hospital Luis Lagomaggiore, Mendoza
  - Hospital Papa Francisco, Salta
  - Hospital San Bernardo, Salta

IPD SHARING:
Plan to Share IPD: Undecided